CLINICAL TRIAL: NCT03594968
Title: Polycystic Ovary Syndrome With Periodontal Disease and Dental Caries
Brief Title: Oxidative Stress in Polycystic Ovary Syndrome With Periodontal Disease and Dental Caries Lesions
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gul Yildiz Telatar, Assistant Professor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 40986104-799
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Polycystic Ovary Syndrome; Dental Caries
MeSH Terms: conditions — Polycystic Ovary Syndrome; Dental Caries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- polycystic ovary syndrome (PCOS): Presence of ≥2 of the following:
  1. oligomenorrhea and/or anovulation
  2. Hyperandrogenism (clinical and/or biochemical) One of the signs for clinical hyperandrogenism is hirsutism, which represents hair growth in a male pattern on a female with four different degrees of severity in 11 different body parts: 1) upper lip; 2) chin; 3) chest; 4) upper back; 5) lower back; 6) upper abdomen; 7) lower abdomen; 8) arm; 9) forearm; 10) thigh; and 11) lower leg. The Ferriman-Gallwey scoring system is used to score the degree of excess male-pattern body hair to indicate hirsutism.
  Interventions: Diagnostic Test: polycystic ovary syndrome
- healthy: healthy patients who had no polycystic ovary
  Interventions: Diagnostic Test: polycystic ovary syndrome

INTERVENTIONS:
Diagnostic Test: polycystic ovary syndrome — 3 to 5th day of the women's normal cycle, we will perform a routine gynecological examination, a basic vaginal ultrasound, a basal hormone profile evaluation
  Other Names: [LH],; [total T],; [free T],; [DHEA-S],; 17-OH-progesterone; [FSH],

SUMMARY:
This study evaluates the oxidative stress parameters in females with polycystic ovary syndrome (PCOS) and clinically healthy. Because of the fact that both oral disease included periodontitis and dental caries, and metabolic syndrome are associated with systemic inflammation, these two disorders may be linked through a common pathophysiologic pathway

DETAILED DESCRIPTION:
Power analysis was performed with the G-Power software package to determine sample size. To cover possible data loss, 10% of a group were added to each group. Medical and dental examination will be performed both of control and experimental groups. Age and body mass index (BMI) will be recorded.

In dental examination decayed, missing, or filled teeth (DMFT) index will be used according to World Health Organization (WHO 1997) criteria. All teeth were visually using the International Caries Detection and Assessment System (ICDAS-II). To analyze the correlation between oral health status and polycystic ovary syndrome linear regression test and for comparison of both the groups (case and control), two sample t test and chi square test were used.

ELIGIBILITY:
Inclusion Criteria:

* females with Polycystic Ovary Syndrome

Exclusion Criteria:

* history of ovarian surgery, patients with thyroid or prolactin hormone level abnormalities, non-classic 21-hydroxylase deficiency and hormonal therapy, steroid drug use past 6 months, obese patients (body mass index, BMI > 35), acute or chronic upper respiratory tract diseases, dental fluorosis, patients using fluoride supplements or orthodontic appliances will not be included in the study.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients were aged from 18 to 24 years, 206 females
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
FSH hormone ovarian morphology (PCOM) | 1 Day
  follicle-stimulating hormone [FSH] is tested by blood sample 6.3_24 mlu/ml
luteinizing hormone | 1 day
  luteinizing hormone [LH] is tested by blood sample 1.68-15 U/L
dehydroepiandrosterone-sulfate | 1 day
  dehydroepiandrosterone-sulfate [DHEA-S] is tested by blood sample 65 to 380 µg/dL or 1.75 to 10.26 µmol/L
17-OH-progesterone | 1 day
  17-OH-progesterone is tested by blood sample 20-100 ng/dL

SECONDARY OUTCOMES:
dental examination | 1 Day
  All teeth were visually using the International Caries Detection and Assessment System (ICDAS-II). The chosen sites were recorded as: 0 = sound;
  1. = first visible sign of noncavitated lesion seen only when the tooth is dried;
  2. = visible noncavitated lesion seen when wet and dry;
  3. = microcavitation in enamel;
  4. = noncavitated lesion extending into dentine seen as an undermining shadow;
  5. = small cavitated lesion with visible dentine: less than 50% of surface;
  6. = large cavitated lesions with visible dentine in more than 50% of the surface.
periodontal examination | 1 Day
  A single calibrated examiner measured probing depth-PD, 0: healthy
  bleeding calculus 3:3.5-5.5 mm 4: over 5.5 mm
Clinical attachment level | 1 Day
  A single calibrated examiner measured clinical attachment level- CAL, 0: 0-3 mm 1:4-5 mm 2:6-8 mm 3:over 8mm 4: 9-11 mm 5: over 12 mm
Plaque Examination | 1 Day
  The plaque amount is scored by using Silness&Löe Plaque Index Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3.
  0:no plaque
  1. A film of plaque
  2. soft deposit s within the gingival pocket
  3. Abundance of soft matter within the gingival pocket.
  Calculation: Total scores of 6 (16, 12, 24, 36, 32, 44) teeth / No of surfaces examined
  Healthy = PI<0.4. Mild = PI 0.4-1.0. Moderate = PI 1.1-2. Severe = PI>2.
Gingival Examination | 1 Day
  0= Normal gingiva;
  1. Mild inflammation
  2. Moderate inflammation
  3. Severe inflammation Calculation: Total scores/ no of surfaces examined 0.1-1:Mild gingivitis, 1.1-2:moderate gingivitis; 2.1-3:severe gingivitis
Bleeding Examination | 1 Day
  0: no bleeding
  1: bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Gül Yıldız Telatar, Principal Investigator — Recep Tayyip Erdogan University Dentistry Faculty
Locations (1):
- Recep Tayyip Erdogan University, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will be available within 6 months of study finishing

REFERENCES:
- [Background] Ozcaka O, Ceyhan BO, Akcali A, Bicakci N, Lappin DF, Buduneli N. Is there an interaction between polycystic ovary syndrome and gingival inflammation? J Periodontol. 2012 Dec;83(12):1529-37. doi: 10.1902/jop.2012.110588. Epub 2012 Apr 17. PMID 22509751
- See also: Polycystic Ovary Syndrome and Gingival Inflammation — http://www.ncbi.nlm.nih.gov/pubmed/22509751